CLINICAL TRIAL: NCT04670198
Title: A Randomised Waiting-list Feasibility Study and Process Evaluation of a Psychosocial Education Programme for Young People With Type 1 Diabetes - the Youth Empowerment Skills (YES)
Brief Title: A Psychosocial Education Programme for Young People With Type 1 Diabetes - the Youth Empowerment Skills (YES)
Acronym: YES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: D-UK 19/0006055
Record Dates: First submitted 2020-11-17; First posted 2020-12-17 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Adolescent; Psychosocial Support Systems
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The study has been designed as a waiting-list randomised controlled trial (RCT). Young people will be randomised to either the phase 1 YES group or the waiting-list control group. The phase 1 YES group will then attend the programme, both groups will be followed-up initially for 6 months, at which point the waiting-list control participants will attend the YES programme in phase 2. Both groups will then be followed-up for a further 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive the Youth Empowerment Skills (YES) programme.
  Interventions: Behavioral: Youth Empowerment Skills
- Waiting-list control (Other): The waiting-list control arm will receive usual care for six months before receiving the Youth Empowerment Skills (YES) programme.
  Interventions: Behavioral: Waiting-list control

INTERVENTIONS:
Behavioral: Youth Empowerment Skills — The Youth Empowerment Skills (YES) programme is a novel psychoeducational intervention with simulation-based experiential learning tailored to the needs of young people. It is based on a social-cognitive learning model, and comprises attendance at 3 all-day YES sessions in non-healthcare settings (groups of 10); and then post-programme networking through social media and follow-up events facilitated by the youth worker. Sessions are led by a peer-educator and a health professional
  Arms: Intervention
Behavioral: Waiting-list control — Usual care for 6 months, followed by the YES programme.
  Arms: Waiting-list control

SUMMARY:
Adolescence is a period of intense physiological, psychological and social change. It can be a challenging period for young people with Type 1 diabetes and is associated with worsening blood sugar control and care disengagement. The investigators have co-designed with young people a psychologically modelled educational programme - Youth Empowerment Skills (YES), which aims to facilitate a positive adaption to living with diabetes while improving knowledge and self-management behaviours. Integrated programme components include social and peer-based learning, immersive simulations, and an outreach youth worker.

The aim of this study is to test the feasibility of the YES programme (acceptance, implementability, recruitment and completion), and estimate its efficacy in relation to metabolic and psychosocial outcomes. The investigators will recruit young people with Type 1 diabetes and conduct a feasibility randomised controlled trial (waiting-list design) with integrated process evaluation. Sixty young people will be randomised to either YES intervention or waiting-list control and evaluate outcomes at 6-months; at this point the waiting list participants will be offered the YES intervention with further follow-up at 12 months.

DETAILED DESCRIPTION:
The study has been designed as a feasibility study with an integrated process evaluation following MRC guidance (Craig et al., 2008; Moore et al., 2015). The process evaluation data collection has been modelled on the COM_B and the Behaviour Change Wheel framework (BCW) frameworks (Michie et al., 2014; Barker et al., 2016) addressing: policy context; intervention functions; target behaviours; and outcomes. As part of the process evaluation the investigators will also use Consolidated Framework for Implementation Research (CFIR) to study how the programme can be optimally embedded within routine diabetes care, and to optimise the design of a subsequent trial (Murray et al., 2010). The investigators will conduct a feasibility randomised controlled trial (waiting-list design) with integrated process evaluation designed following the Medical Research Council's (MRC) Complex Intervention Evaluation Framework (Craig et al., 2008). Sixty young people will be randomised to either YES intervention or waiting-list control and evaluate outcomes at 6-months; at this point the waiting list participants will be offered the YES intervention with further follow-up at 12 months.

The proportion of patients achieving the progression criteria and the target reduction in glycated haemoglobin (HbA1c) from baseline to follow-up (6 and 12 months) will be estimated in both intervention and waiting list control groups. The investigators will also estimate the standard deviation (SD) of the mean difference between the intervention and waiting list control groups in HbA1c at 6 and 12 months. These statistics will help to inform the sample size calculation of a larger trial.

The process evaluation will consider the setting, implementation, and mechanisms of action of the programme to support interpretation of the outcomes. The process evaluation uses a standardised taxonomy for understanding implementation (Julious, 2005; Proctor et al., 2011), and will assess: the reach, fidelity and receipt of the programme; acceptability, appropriateness and feasibility; unintended consequences; potential sustainability; and implementation costs and strategies. In addition, potential mechanisms of action will be elicited, including changes in behaviours, and how they relate to programme delivery and outcomes.

The investigators will use a mixed-method approach with validated implementation outcome surveys (Powell et al., 2015) and one-to-one interviews with young people, their relatives and healthcare professionals. The data collection tools and analytic models have been designed with reference to the BCW (Michie et al., 2014) and to provide the data for CFIR analysis, considering the barriers and facilitators to the intervention. To ensure relevance and feasibility, the data collection procedures will be refined with the study patient and public involvement groups. Data collection will be conducted at multiple time points to provide opportunities for data triangulation and subsequent theory generation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 diabetes
* Sub-optimal glycaemic control (HbA1c 8.5%)
* No current or planned attendance at other structured education programmes

Exclusion Criteria:

* Severe, physical/mental illness
* Pregnancy
* Unstable retinopathy
* Significant learning difficulties

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | Baseline, 6 months, 12 months
  HbA1c will be used to measure:
  1. the number of participants achieving clinically significant reductions of 5.5mmol/mol or more and mean differences between groups over time
  2. the standard deviation (SD) of the mean difference between the intervention and control group in HbA1c at 6 months; for the control group the SD of the mean difference between HbA1c at 12 months and pre-exposure (phase 2) and for the phase 1 intervention group the SD of the mean HbA1c difference between post (6 and 12 months) and pre-exposure.

SECONDARY OUTCOMES:
Frequency of blood glucose monitoring | Baseline, 6 months, 12 months
  Participants' glucose meters will be downloaded to assess the number of participants with 20% increase in frequency of glucose monitoring between pre- and post-intervention exposure, and any difference between intervention and control groups at 6 months.
Insulin adherence | Baseline, 6 months, 12 months
  Insulin adherence will be measured by self-report scale to assess the number of participants reporting a change in insulin adherence between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months.
  Maximum score is 10 and minimum score is 2. Higher scores indicate better adherence.
Self-Management of Diabetes in Adolescence Scale (SMOD-A) | Baseline, 6 months, 12 months
  The SMOD-A will be used to assess any change in self-management of diabetes between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months. This consists of five subscales.
  Subscale 1: Collaboration with Parents. The range of scores is 0 to 39. Higher scores indicate more collaboration.
  Subscale 2: Diabetes Care Activities. The range it 0 to 45. Higher scores indicate more/better performance of these diabetes tasks.
  Subscale 3: Diabetes Problem-Solving. Range of scores is 0 to 21. Higher scores indicate better/more problem-solving.
  Subscale 4: Diabetes Communication. The range of scores is 0 to 30. Higher scores indicate better/more communication.
  Subscale 5: Goals. The range of scores is 0 to 21. Higher scores indicate more goals.
Confidence in Diabetes Self-Care Scale (CDSS) | Baseline, 6 months, 12 months
  The CDSS will be used to measure any change in confidence in diabetes self-care between pre-and post-intervention exposure, and between intervention and control groups at 6 months. Maximum value is 100, minimum value is 20. Higher score means more confidence.
Diabetes Quality of Life Instrument (DQOL) (adapted for youth) | Baseline, 6 months, 12 months
  The DQOL will be used to assess any change in quality of life between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months.
  DQOL has 3 subscales:
  Subscale 1: Impact of diabetes. Maximum value is 120. Minimum value is 24. Higher scores indicate more impact of diabetes on quality of life.
  Sunscale 2: Worries about diabetes. Maximum score is 55. Minimum score is 11. Higher scores mean more worries.
  Subscale 3: Satisfaction with life. Maximum score 85. Minimum score 5. Higher score means more satisfied.
Brief Illness Perception Questionnaire (IPQ-B) | Baseline, 6 months, 12 months
  The IPQ-B will be used to measure any change in diabetes perception between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months. Each of the eight dimensions measured uses a maximum score of 10 and a minimum score of 0. A higher score indicates more severe perception of illness.
Emergency care events | Baseline, 6 months, 12 months
  The number of ambulance call-outs, Accident & Emergency attendance and hospitalisations will be taken from hospital records to assess any change in number of events between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months.
Hypoglycaemia and severe hypoglycaemic events | Baseline, 6 months, 12 months
  Hypoglycaemia is defined as blood glucose 3.5 mmol/L and severe hypoglycaemic events are defined as requiring 3rd party assistance. The number of events will be taken from hospital records to assess any change in hypoglycaemia and severe hypoglycaemic events between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months.
Weight | Baseline, 6 months, 12 months
  Participants will be weighed at baseline, 6 and 12 months to assess any change in weight between pre- and post-intervention exposure, and the difference between intervention and control groups at 6 months.
Intervention Appropriateness Measure (IAM) | Within 3 months of intervention
  Intervention Appropriateness Measure will be used to assess the appropriateness of the intervention. It is a four-item questionnaire measuring implementation outcomes. Score values range from 1 to 5. The higher the score the more appropriate the intervention.
Feasibility of Intervention Measure (FIM) | Within 3 months of intervention
  Feasibility of Intervention Measure will be used to assess the feasibility of the intervention. It is a four-item questionnaire measuring implementation outcomes. Score values range from 1 to 5. The higher the score the more feasible the intervention.
Acceptability of Intervention Measure (AIM) | Within 3 months of intervention
  Acceptability of Intervention Measure will be used to assess the acceptability of the intervention. It is a four-item questionnaire measuring implementation outcomes. Score values range from 1 to 5. The higher the score the more acceptable the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Angus Forbes, Principal Investigator — King's College London
Locations (5):
- United Kingdom (5):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University Lewisham Hospital, London
  - Queen Elizabeth Hospital, London
  - King's College Hospital, London
  - St George's University Hospital HS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available at the end of the study.
Access Criteria: Requests made to study researchers

REFERENCES:
- [Derived] Kariyawasam D, Soukup T, Parsons J, Sevdalis N, Baldellou Lopez M, Forde R, Ismail K, Jones M, Ford-Adams M, Yemane N, Pender S, Thomas S, Murrells T, Silverstien A, Forbes A. Protocol for a feasibility study and process evaluation of a psychosocially modelled diabetes education programme for young people with type 1 diabetes: the Youth Empowerment Skills (YES) programme. BMJ Open. 2022 Jun 9;12(6):e062971. doi: 10.1136/bmjopen-2022-062971. PMID 35680254